CLINICAL TRIAL: NCT07315438
Title: Model-Informed Precision Dosing on Amikacin and Vancomycin Therapy in Critically Ill Children: A Pilot Randomized Clinical Trial
Brief Title: Model-Informed Precision Dosing on Amikacin and Vancomycin Therapy in Critically Ill Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nadir Yalçın, Director, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neo-MIPD
Record Dates: First submitted 2025-11-28; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Model Informed Precision Dosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIPD Group (Experimental)
  Interventions: Device: MIPD Tool
- Standard of Care Group (No Intervention)

INTERVENTIONS:
Device: MIPD Tool — It is a precision dosing platform that combines population pharmacokinetic/pharmacodynamic (popPK/PD) modeling with artificial intelligence and machine learning to optimize individualized drug therapy.
  It uses patient-specific demographic, clinical, and laboratory data to generate real-time personalized dosing recommendations based on validated popPK models.
  Arms: MIPD Group

SUMMARY:
Achieving optimal antibiotic exposure in critically ill pediatric patients is difficult due to (their) dynamic physiology and variability. Conventional weight-based regimens often fail to reach pharmacokinetic/pharmacodynamic (PK/PD) targets for narrow therapeutic index agents such as vancomycin and amikacin. Model-Informed Precision Dosing (MIPD), which integrates Bayesian forecasting with population pharmacokinetics (popPK), offers a potentially valuable yet underexplored approach in pediatric intensive care to better attain and sustain target exposure. This pilot randomized clinical trial evaluated MIPD-guided dosing of vancomycin and amikacin using InsightRX Nova® versus standard of care (SoC) in a tertiary PICU. Patients whose model-recommended doses matched standard regimens were analyzed under SoC. Primary outcomes included prediction accuracy (a priori vs a posteriori) and model fit; secondary outcomes assessed dose optimization, inflammatory response, renal safety, treatment duration, and mortality.

ELIGIBILITY:
Inclusion Criteria

* Hospitalized patients (NICU) receiving vancomycin or amikacin
* Treatment with vancomycin or amikacin initiated during hospitalization
* At least one therapeutic drug monitoring (TDM) measurement obtained Exclusion Criteria
* Failure to obtain written informed consent
* Death within the first 24 hours after treatment initiation
* Discontinuation of therapy before the first TDM measurement
* Determined unsuitable for study participation by the treating physician

Ages: 38 Months to 81 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Predictive Accuracy of Model-Informed Precision Dosing (MIPD) Based on Median Absolute Error (MdAE) | From first therapeutic drug monitoring (TDM) sample to second TDM sample (typically within 3-5 days of therapy)
  Predictive accuracy of the pharmacokinetic model will be evaluated by calculating the Median Absolute Error (MdAE) between model-predicted and observed antibiotic serum concentrations. MdAE was prespecified as the primary accuracy metric due to its robustness to outliers in small pediatric samples.
Predictive Accuracy of Model-Informed Precision Dosing (MIPD) Based on Mean Absolute Error (MAE) | From first therapeutic drug monitoring (TDM) sample to second TDM sample (typically within 3-5 days of therapy)
  Mean Absolute Error (MAE) between model-predicted and observed serum antibiotic concentrations will be calculated to assess overall prediction error.
Predictive Accuracy of Model-Informed Precision Dosing (MIPD) Based on Median Error (MdE) | From first therapeutic drug monitoring (TDM) sample to second TDM sample (typically within 3-5 days of therapy)
  Median Error (MdE) will be calculated to evaluate directional bias between predicted and observed serum antibiotic concentrations.

SECONDARY OUTCOMES:
Change in C-Reactive Protein (CRP) Level | Baseline to approximately day 3-5 of therapy
  The absolute change in serum C-reactive protein (CRP) level from baseline (within 24 hours of antibiotic initiation) to the time of the second TDM sample will be evaluated as an inflammatory response marker.
Change in Procalcitonin Level | Baseline to approximately day 3-5 of therapy
  The absolute change in serum procalcitonin level from baseline to the time of the second TDM sample will be assessed.
Change in Serum Creatinine Level | Baseline to approximately day 3-5 of therapy
  The absolute change in serum creatinine level from baseline to the time of the second TDM sample will be evaluated as a marker of renal safety.
Change in Pharmacokinetic Model-Fit Category | From first to second TDM sample (typically within 3-5 days)
  Within-patient change in pharmacokinetic model-fit category (poor, intermediate, good) between the first and second TDM measurements will be assessed to evaluate improvement in model performance after Bayesian updating.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No